CLINICAL TRIAL: NCT04252222
Title: The VL3 Videolaryngoscope for Elective Tracheal Intubation in Adults: a Prospective Pilot Study
Brief Title: The VL3 Videolaryngoscope for Elective Tracheal Intubation in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Giuseppe Pascarella, Medical Doctor, Unit of Anesthesia and Intensive Care, Campus Bio-Medico University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 82/18 OSS ComET CBM
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Difficult Airway Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VL3 (Experimental): Tracheal intubation with VL3 videolaryngoscope
  Interventions: Device: Videolaryngoscopy with VL3

INTERVENTIONS:
Device: Videolaryngoscopy with VL3 — Tracheal Intubation aided by VL3 Videolaryngoscope

SUMMARY:
We conducted an observational prospective pilot study to assess the efficacy of the VL3 videolaryngoscope for routinely tracheal intubation in 56 adults, in terms of successful rate, no. attempts and manoeuvre duration, including both normal and difficult airways.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidates for general anesthesia in elective surgery
* Age over 18 years
* ASA physical status I-III.

Exclusion Criteria:

* Paediatric population
* ASA physical status IV
* Emergency tracheal intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Tracheal intubation rate | 30 minutes
  successful tracheal intubation rate using VL3 video laryngoscope
Number of attempts | 30 minutes
  Number of attempts for a successful tracheal intubation
Total time of intubation | 15 minutes
  Time needed to perform a tracheal intubation from the insertion of VL3 video laryngoscope into the patient mouth
Time to glottis visualization | 15 minutes
  Time needed to visualize the glottis from the insertion of VL3 video laryngoscope into the patient mouth
Cormack-Lehane grade | 15 minutes
  Cormack-Lehane grade observed at videolaryngoscopy

SECONDARY OUTCOMES:
Need for external laryngeal pressure | 15 minutes
  Need for external laryngeal pressure during laryngoscopy
Presence of post-laryngoscopy side effects | 3 days
  Presence of post-laryngoscopy side effects (bleeding, postoperative sore throat and/or dysphonia)

CONTACTS AND LOCATIONS:
Locations (1):
- Università Campus Biomedico, Roma, Italy

IPD SHARING:
Plan to Share IPD: No